CLINICAL TRIAL: NCT05670184
Title: The Effect of LSD on Neural Synchrony, Prosocial Behavior, and Relationship Quality
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: NL80435.068.22
Record Dates: First submitted 2022-11-30; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-11

CONDITIONS: Prosocial Behavior
MeSH Terms: conditions — Altruism | interventions — Lysergic Acid Diethylamide; Ethanol

STUDY DESIGN:
Intervention Model Description: LSD and placebo will be administered in an AB or BA sequence, with half of the couples following sequence AB and the other half following sequence BA. Couples will receive an oral dose of either 50 µg of LSD or placebo. All couples will receive both the LSD and the placebo solution on separate dosing days with follow-ups 2 days later (in the lab), and 4 days later (at home). There will be a 14-day washout period between drug administrations.
Who Masked: Participant, Investigator
Masking Description: Random allocation of couples to a the treatment order will be done using Sealedenvelope software, by one experimenter who does not come in direct contact with the participants. The study will be double blind to the subject and the testing experimenter. One experimenter will be responsible for preparing the LSD. This experimenter will not be the one testing the participants. If a subject is withdrawn from the study they will be replaced, for a maximum of n=60 participants (n=30 couples). Following completion of all data collection the study will be fully unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LSD condition (Experimental): 60 participants will receive LSD.
  Interventions: Drug: LSD
- Ethanol condition (Placebo Comparator): 60 participants will receive placebo.
  Interventions: Drug: Ethanol

INTERVENTIONS:
Drug: LSD — Single dose of LSD (50 µg) will be administered in a small amount of alcohol (ethanol, 2ml/95% Vol.) orally.
  Other Names: lysergic acid diethylamide
  Arms: LSD condition
Drug: Ethanol — Identical ampules containing pure ethanol without the investigational product will be used (1mL ethanol, 95% Vol.).
  Arms: Ethanol condition

SUMMARY:
The goal of this study is to assess the effects of LSD on neural synchrony, prosocial behavior, and relationship quality in healthy romantic couples.

DETAILED DESCRIPTION:
Evidence is growing that psychedelic substances such as psilocybin, lysergic acid diethylamide (LSD) and ayahuasca could be a potential alternative treatment option for common and difficult to treat psychiatric conditions. One proposed mechanism that psychedelics target, which is a hallmark of seemingly all psychiatric disorders, are deficits in social cognitive abilities. However, the neural underpinnings of psychedelic induced alterations in prosocial behavior are currently unknown. The investigators hypothesize psychedelics increase such prosocial behaviors by increasing neural synchrony, which is the coupling of brain-to-brain activity across two or more people; it has been found to underlie social connection and various forms of shared prosocial behavior.

The current project will primarily assess whether LSD enhances neural synchrony between romantic partners. Second, the investigators will assess whether LSD enhances prosocial behavior between members of a dyad, thus replicating previous studies which assessed prosocial behavior within one individual at a time. The investigators will also assess the relationship between neural synchrony and outcome variables of the prosocial behaviour tasks. Lastly, it will be assessed whether LSD-induced changes in neural synchrony and/or prosocial behaviour affect persisting relationship quality. Oxytocin and cytokine concentrations, will also be quantified to investigate whether there is a relationship between these factors and changes in prosocial behaviour.

The study design will be conducted according to a double-blind, placebo-controlled, 2-way crossover design. Healthy participants (N=60) who are in a relationship (N=30 couples) will receive placebo and an oral dose of 50 µg of LSD. Between each condition, there will be a minimum of 14 days washout. This leads to a total study duration of minimally four weeks, for a participant to go through the medical examination and both drug conditions.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Understanding the procedures and the risks associated with the study.
* Age between 18 and 35 years old.
* Being in a steady relationship for at least 6 months.
* Proficient knowledge of the English language
* Previous experience with at least one psychedelic drug (psilocybin, LSD, mescaline, Ayahuasca, DMT, 5-MeO-DMT), but not within the past 3 months
* Absence of any major medical condition as determined by medical examination and laboratory analysis
* Absence of any major psychological condition as determined by medical examination
* Free from psychotropic medication
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no coffee, black or green tea, or energy drink after midnight of the evening before the study session, as well as during the study day.
* Participants must be willing not to drive a traffic vehicle or to operate machines within 24 h after substance administration.
* Normal weight, body mass index (weight/height2) between 18 and 28 kg/m2

Exclusion Criteria:

* History of drug addiction (determined by the medical questionnaire, drug questionnaire and medical examination)
* Previous experience of serious side effects to psychedelic drugs (anxiety or panic attacks)
* Pregnancy or lactation
* Hypertension (diastolic > 90 mmHg; systolic > 140 mmHg)
* Current or history of psychiatric disorder (determined by the medical questionnaire and medical examination)
* Psychotic disorder in first-degree relatives
* Any chronic or acute medical condition
* History of cardiac dysfunctions (arrhythmia, ischemic heart disease,…)
* For women: no use of a reliable contraceptive
* Tobacco smoking (>20 per day)
* Excessive drinking (>20 alcoholic consumptions per week)
* Experience with a full dose of a psychedelic within the last three months
* Current use of SSRI medication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Neural synchrony | On the acute dosing test day, 1.5-2 hours after substance administration
  Quantification of neural synchrony between members of a couple utilizing previously validated naturalistic interaction paradigms, including a motor cooperation task, empathy giving task, and affective touch and eye contact paradigm, will be employed. Resting state EEG will be used as a control.

SECONDARY OUTCOMES:
Empathy | On the acute dosing test day, 2 hours (EGT) and 3 hours (MET) after substance administration
  Cognitive and emotional empathy will be assessed via the empathy giving task (EGT) and the multifaceted empathy test (MET).
Self-other distinction | On the acute dosing day, 2.5 hours (SMS) after substance administration. The OIS will be administered repeatedly at baseline (-0.5 hours), 2 hours, 3 hours, 4.5 hours, and 7 hours after substance administration, and at 2 days follow up.
  The degree of self-other merging will be assessed using synchronous multisensory stimulation (SMS), and responses on the inclusion of other in the self scale (OIS).
Prosocial behavior | On the acute dosing day, 6 hours after substance administration. The PET will also be administered at 2 days follow-up.
  Prosocial behavior will be assessed via participants' response rate on the prosocial learning task (PLT), and the amount of effort for other individual in the prosocial effort task (PET).
Social influence processing | On the acute dosing day, 3 hours after substance administration
  Social influence processing will be assessed via participants' degree of rating adjustment after feedback in the social influence paradigm (SIP).
Trust | On the acute dosing day, 6.5 hours after substance administration
  The trust game for couples (TGC) will assess participants' willingness to invest personal resources in pro-relationship attitudes.
Creativity | On the acute dosing day, 5.5 hours (CFO, PST) after substance administration. The DAT will be administered at 2 days follow-up.
  Creativity will be assessed by the semantic distance in the chain free association (CFO) and the divergent association tasks (DAT), and also by the ability to separate old and new information in the pattern separation task (PST).
Sociality | On the acute dosing day, SRQ will be administered at 4.5 hours after substance administration, while the VAS-S will be administered at baseline (-0.5 hours), at 1, 2, 3, 4, 5, 6, and 7 hours after substance administration.
  Sociality will be measured by the social reward questionnaire (SRQ) and the visual analogue scales that measure feelings of social behavior (VAS-S).
Conflict resolution | At 2 days follow-up.
  The couples conflict resolution (CR) task will measure the duration of positive and negative behavior of members of a couple via video recordings of couples' interactions.

OTHER OUTCOMES:
Relationship quality | At baseline, 2 days follow-up (CSI) and at 4 days follow-up (CSI, PPRS, ECR, IRI-C).
  Relationship quality will be measured via subjective reports on a number of scales: the couples satisfaction index (CSI), the perceived partners responsiveness scale (PPRS), the experiences in close relationship scale (ECR), and the interpersonal reactivity index for couples (IRI-C).
Sexual function | At baseline, 2 days follow-up (GMSEX), and at 4 days follow-up (GMSEX, FSFI/IIEF).
  Sexual function will be measured via subjective reports on a number of scales: the global measure of sexual satisfaction (GMSEX), the female sexual function index (FSFI), and the international index of erectile function (IIEF).
Well-being | On the acute dosing day, at baseline (-0.5 hours) and at 7 hours after substance administration, at the 2 day follow-up, and at the 4 day follow-up.
  Well-being will be measured via subjective reports on the satisfaction with life scale (SWLS).
Subjective drug effects | On the acute dosing day, 7 hours after substance administration.
  Subjective drug effects will be measured via subjective reports on the altered states of consciousness rating scale (5D-ASC), and on the ego dissolution inventory (EDI).
Real-time social behavior | Daily up until 3 days after the acute dosing day.
  Real-time social behavior will be assessed via subjective reports on experience sampling questions (ESQ) in the Ethica app.
LSD concentrations | Acute dosing day:baseline (-0.5 hour), at 1.5, 2.5, 3.5, 5, and at 7 hours.
  Blood samples will be collected to measure LSD concentrations
Oxytocin concentrations | Acute dosing day:baseline (-0.5 hour), at 1.5, 2.5, 3.5, and 4.5 hours after substance administration.
  Blood samples will be collected to measure oxytocin
Metabolomics concentration | Acute dosing day:baseline (-0.5 hour), at 1.5 and 7 hours after substance administration.
  Blood samples will be collected to measure metabolomics
Inflammatory cytokines | Acute dosing day:baseline (-0.5 hour), at 1.5 hours and 2 days after substance administration.
  Blood samples will be collected to measure inflammatory cytokine levels
Aftercare | At the end of the 2 day followup
  Any lasting negative effects of the drug will be assessed via a visual analogue scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Johannes G Ramaekers, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands